CLINICAL TRIAL: NCT03463408
Title: Pilot Study of Neoadjuvant Dual Checkpoint Blockade With Concurrent Radiation in Resectable Soft Tissue Sarcoma
Brief Title: Immunotherapy + Radiation in Resectable Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Adrienne Victor, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USAR17101
Record Dates: First submitted 2017-12-24; First posted 2018-03-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma
Keywords: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: two cohort, open label, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunotherapy arm (Experimental): Cohort A will comprise adult soft tissue sarcoma patents who consent to and receive ipilimumab + nivolumab concurrently with standard of care radiation. Ipilimumab will be given at a dose of 1 mg/kg every 6 weeks (total two doses) and nivolumab given as a flat dose of 240 mg every 2 weeks (total four doses).
  Standard surgical resection will be done 2 to 4 weeks after completion of radiotherapy. Accrual is expected to occur over 2 years. Follow up data will be collected for up to 3 years post-treatment.
  Interventions: Drug: nivolumab; Drug: ipilimumab
- no immunotherapy arm (No Intervention): Cohort B will comprise patients eligible for the trial who do not wish to receive immunotherapy but consent to the same blood draws, surveys, and specimen analysis as Cohort A. Cohort B will serve as a non-randomized but pragmatic and clinically relevant control group.
  Standard surgical resection will be done 2 to 4 weeks after completion of radiotherapy. Accrual is expected to occur over 2 years. Follow up data will be collected for up to 3 years post-treatment.

INTERVENTIONS:
Drug: nivolumab — 240 mg every 2 weeks
  Arms: Immunotherapy arm
Drug: ipilimumab — 1 mg/kg every 6 weeks
  Arms: Immunotherapy arm

SUMMARY:
Immunotherapy + Radiation in Resectable Soft Tissue Sarcoma

DETAILED DESCRIPTION:
A single institution two cohort, open label, non-randomized study of neoadjuvant nivolumab and ipilimumab with concurrent radiation followed by surgical resection.

Cohort A will comprise adult soft tissue sarcoma patents who consent to and receive ipilimumab + nivolumab concurrently with standard of care radiation. Ipilimumab will be given at a dose of 1 mg/kg every 6 weeks (total two doses) and nivolumab given as a flat dose of 240 mg every 2 weeks (total four doses).

Cohort B will comprise patients eligible for the trial who do not wish to receive immunotherapy but consent to the same blood draws, surveys, and specimen analysis as Cohort A. Cohort B will serve as a non-randomized but pragmatic and clinically relevant control group.

Peripheral blood will be collected on day 1 pre-treatment, day 14, day 42, immediately prior to surgery, and at 3 month follow up. Peripheral blood will be sent for multidimensional flow analysis of changes in immune cell composition and markers of proliferation. Serum samples will be obtained before starting treatment and after surgery. Samples from select subjects whose resected tumors show significant response and whose tumors showed minimal response will be sent to Serametrix for serum profiling to detect antibody response to a panel of tumor-specific antigens.

Standard surgical resection will be done 2 to 4 weeks after completion of radiotherapy. Accrual is expected to occur over 2 years. Follow up data will be collected for up to 3 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with biopsy-proven soft-tissue sarcoma with confirmatory pathology review at University of Rochester Medical Center (URMC)
* 18 years or older.
* Able to provide informed consent.
* Resectable disease per surgical evaluation.
* Neoadjuvant/preoperative radiotherapy has been recommended
* Intermediate to high grade sarcoma on biopsy, tumor > 5 cm in size by imaging
* Willing to have blood draws for flow cytometry and Serametrix analysis.
* Willing to receive neoadjuvant radiation therapy and subsequent surgical resection.
* Patients with known human immunodeficiency virus (HIV) are eligible if the lymphocytes > 350 CD4+ cells and no detectable viral load.
* Women of childbearing potential (defined as any woman, who 1) has not undergone tubal ligation, a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months or has had menses at any time in the preceding 24 consecutive months):

  * Must not be pregnant or nursing
  * Must have a negative pregnancy test done within 7 days prior to registration as well as within 72 hrs. prior to receiving first dose of study medication
  * Women of childbearing potential must use at least two other accepted and highly-effective methods of contraception and/or agree to abstain from sexual intercourse for at least 5 months after the last dose of nivolumab and/or ipilimumab.
  * Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Sexually active males must use at least two other accepted and highly-effective methods of contraception and/or agree to abstain from sexual intercourse for at least 7 months after the last dose of nivolumab and/or ipilimumab
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2

Exclusion Criteria:

* Gastrointestinal stromal tumor, dermatofibrosarcoma protuberans, rhabdomyosarcoma, Ewing's sarcoma, low-grade sarcomas, osteosarcoma subtypes
* History of radiation to the affected area
* Evidence of metastatic disease prior to treatment
* Any history of prior therapy with ipilimumab or nivolumab, or any agent targeting PD-1, PD-L1 or CTLA-4.
* History of any the following:

  * Active known or suspected autoimmune disease
  * Active autoimmune colitis
  * Autoimmune pan hypopituitarism
  * Autoimmune adrenal insufficiency
  * Known active hepatitis B or C
  * Known active pulmonary disease with hypoxia defined as:
* Oxygen saturation < 85% on room air or
* Oxygen saturation < 88% despite supplemental oxygen
* No systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration.
* Second active malignancy, not including localized basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast; patients with a history of other malignancies are eligible if they have been continuously disease-free for > 3 years prior to the time of registration.
* Absolute neutrophil count (ANC) <= 1,500/mm^3
* Platelet count <= 100,000/mm^3
* AST (Aspartate Aminotransferase) or ALT (Alanine Aminotransferase) => 2 x upper limit of normal (ULN)
* Thyroid stimulating hormone (TSH) outside of normal limits; supplementation is acceptable to achieve a TSH within normal limits; in patients with abnormal TSH if free T4 is normal and patient is clinically euthyroid, patient is eligible.
* Life expectancy under 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event evaluation | 2 years
  Evaluate safety through assessment of adverse events throughout the course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353